CLINICAL TRIAL: NCT06984042
Title: Improving Pain Management in Nursing Homes: A Research Project to Enhance Care Practices
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0084_GERIATRIE
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Pain Management; Nursing Homes; Elderly; Pain; Health Care Quality, Access, and Evaluation; Patient-Centered Care
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Residents of EHPAD: 2 residents
- Family or close: 2 family members or close
- Healthcare professionals: 1 psychologist, 1 head of department, 1 health manager, 2 IDE, 2 AS, 2 AVS and 1 quality engineer.

SUMMARY:
This study aims to improve the way pain is managed in nursing homes. It focuses on training staff, creating better systems to track pain, and involving residents and their families in decision-making. The goal is to provide better, more personalized care for residents, making sure their pain is properly managed and that the staff is well-equipped to support them.

ELIGIBILITY:
Inclusion Criteria

For residents:

* Aged 60 years or older
* Living in the nursing home (EHPAD) for at least 3 months
* Presence of chronic or acute pain requiring regular management
* Willing to participate in a semi-structured interview
* Provided informed and signed consent to participate in the study

For family members or close relatives:

* Family member or close relative who visits the resident regularly
* Actively involved in the resident's care or support
* Willing to participate in a semi-structured interview
* Provided informed consent to participate in the study

For healthcare professionals:

* Registered nurses (RN), nursing assistants (NA), or support staff (AVS) involved in professional practice analysis groups
* Nurse managers, department heads, psychologists of the nursing home, or the hospital's quality engineer participating in semi-structured interviews
* Voluntary participation with informed and signed consent
* Available to participate in all stages of the project

Exclusion Criteria

For residents:

* Under 60 years of age
* Living in the nursing home for less than 3 months
* Absence of pain requiring regular management
* Cognitive impairment preventing participation in interviews
* Refusal or inability to participate in discussion and exchange sessions
* Unwillingness to take part in a semi-structured interview
* Inability to provide informed and signed consent
* Resident in end-of-life care

For family members or close relatives:

* Family member or relative with infrequent contact with the resident
* Refusal or inability to participate in discussion and exchange sessions
* Refusal to sign informed consent for participation
* Unwillingness to take part in a semi-structured interview

For healthcare professionals:

* Refusal or inability to participate in group discussions or semi-structured interviews
* Refusal to sign informed consent for participation
* Temporary, freelance, or external professionals not part of the regular care team
* Professionals mandated or forced to participate in practice analysis groups
* Unavailable to participate in all stages of the project

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from three main groups associated with nursing homes (EHPADs):
  Residents aged 60 years or older, who have been living in the EHPAD for at least 3 months and are experiencing chronic or acute pain requiring regular management. These residents must be capable of giving informed consent and willing to participate in semi-structured interviews.
  Family members or close relatives of residents, who are regularly involved in the resident's life and support, and who are willing and able to participate in interviews and discussions related to the study.
  Healthcare professionals working in the EHPAD, including registered nurses (IDE), nursing assistants (AS), care support staff (AVS), nurse managers, department heads, psychologists, and quality engineers. Participants must be directly involved in care or organizational activities, and available to take part in the full scope of the study.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of residents with regular documentation of pain assessment in the Electronic Health Record | Over a 4-month study period (from June to October 2024).

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France